CLINICAL TRIAL: NCT06815341
Title: Risk Factors for Sub Mucosal Fibrosis During Achalasia Cardia
Brief Title: Risk Factors for Sub Mucosal Fibrosis During Achalasia Cardia: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Other Study IDs: SMF
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Esophagus Disorder
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Classification for Stasis Esophagitis:

Grade I Grade II Grade III Vascular pattern Obscured Obscured Obscured Mucosal thickening No Yes Yes Ulceration No Yes Yes Nodularity No No Yes

DETAILED DESCRIPTION:
Predictors of Submucosal Fibrosis:

Various factors were analysed for prediction of SMF including age, gender, stasis esophagitis, type of achalasia, duration of disease, lower esophageal sphincter pressure (LESP), height of barium column on barium esophagogram and severity of symptoms (Eckardt score). Esophageal mucosa was graded for the severity of stasis esophagitis (grade I to grade III) based on vascular pattern, mucosal thickening, ulceration and nodularity. SMF was graded (I minimal, II moderate, III severe) according to mucosal lift, difficulty in entry, density of SM fibers, separation of mucosa and muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients (between 18 to 75 years of age) who underwent POEM for achalasia or other esophageal motility disorders.
* Had a diagnosis of esophageal achalasia confirmed by High Resolution Manometry, barium esophagogram.

Exclusion Criteria:

* Patients who underwent treatment other than achalasia
* Lost to follow up patients.
* Incomplete clinical record patients
* Patients not willing to participate in the study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 339 subjects
Sampling Method: Probability Sample
Enrollment: 339 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
The primary aim of the study is to evaluate the predictors for Sub mucosal fibrosis in cases with achalasia cardia. | 100 minutes
  sub mucosal fibres determination in different muscles of esophagus

SECONDARY OUTCOMES:
: To improve the technical outcomes of per oral endoscopy myotomy | 100 minutes
  to know the efficacy of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Nabi Dr Mohammed, MBBS MD, Principal Investigator — AIG Hospitals
Locations (2):
- India (2):
  - Asian institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana
  - Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana